CLINICAL TRIAL: NCT03581357
Title: Mobile Mindfulness Meditation Intervention to Improve the Well-Being of Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bantum-2017-1
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cancer, Other Than Non-melanoma Skin Cancer
Keywords: Previous diagnosis of cancer, completed primary treatment of cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized wait-list control design, such that participants will be randomized to either begin the intervention immediately or after 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control/Waitlist (Anxiety Group) (Active Comparator): Subjects assigned to this arm will not be offered access to the mobile app during the first 8 weeks of their participation. Subjects will be asked to begin using the app eight weeks after randomization. Subjects assigned to this arm will complete a questionnaire at three times points: the beginning after the subject has signed the informed consent form, at the 8 week time point (just before subject begins using the mobile app) and 16 week time point.
  Interventions: Behavioral: Mobile Mindfulness Meditation
- Mindfulness App (Anxiety Group) (Active Comparator): Subjects assigned to this arm will receive mindfulness meditation instructions for 8 consecutive weeks following randomization to this arm. The mobile app contains 14 sessions that subject can participate in at their own pace. Subjects are asked to try and practice mindfulness meditation daily, for a total time of 2 hours per week. Subjects assigned to this arm will complete a questionnaire at three times points: the beginning after the subject has signed the informed consent form, at the 8 week and 16 week time points.
  Interventions: Behavioral: Mobile Mindfulness Meditation
- Control/Waitlist (Neuropathy Group) (Active Comparator): Subjects assigned to this arm will not be offered access to the mobile app during the first 8 weeks of their participation. Subjects will be asked to begin using the app eight weeks after randomization. Subjects assigned to this arm will complete a questionnaire at three times points: the beginning after the subject has signed the informed consent form, at the 8 week time point (just before subject begins using the mobile app) and 16 week time point.
  Interventions: Behavioral: Mindfulness Coach
- Mindfulness App (Neuropathy Group) (Active Comparator): Subjects assigned to this arm will receive mindfulness meditation instructions for 8 consecutive weeks following randomization to this arm. The mobile app contains 14 sessions that subject can participate in at their own pace. Subjects are asked to try and practice mindfulness meditation daily, for a total time of 2 hours per week. Subjects assigned to this arm will complete a questionnaire at three times points: the beginning after the subject has signed the informed consent form, at the 8 week and 16 week time points.
  Interventions: Behavioral: Mindfulness Coach

INTERVENTIONS:
Behavioral: Mobile Mindfulness Meditation — It is hypothesized that participants who are randomized in the app condition will have significantly less anxiety, pain, fatigue, and sleep disturbance than their counterparts in the control condition.
  Arms: Control/Waitlist (Anxiety Group); Mindfulness App (Anxiety Group)
Behavioral: Mindfulness Coach — It is hypothesized that participants who are randomized into treatment condition will have significantly less CIPN, anxiety, and fatigue, and improved anxiety, in comparison to their counterparts in the wait-list control condition.
  Arms: Control/Waitlist (Neuropathy Group); Mindfulness App (Neuropathy Group)

SUMMARY:
Evaluate the impact and satisfaction of Mobile Mindfulness Meditation on anxiety, pain, fatigue, trauma, and sleep in cancer survivors.

DETAILED DESCRIPTION:
Through previous research, mindfulness meditation has been linked to decreases in anxiety, increased pain tolerance, better mood, and improved quality of life, in both healthy and medical populations. Although mindfulness meditation is well promoted both clinically and in the media, finding ways to promote engagement in and fidelity to the intervention, in a format that is accessible for cancer survivors is crucial, as the availability of resources and appreciation of the benefits does not necessarily lead to behavior change.

With many more people surviving cancer than in previous decades, there is an opportunity to act on the residual effects of cancer diagnosis and treatment, and with the prevalence of technology ever increasing, online and mobile interventions have become more frequently delivered and have a particular utility for this population. Physical and geographic limitations could prevent cancer survivors from accessing psychosocial interventions. Whether the repeated beneficial findings of face-to-face training in mindfulness meditation will be found in a mobile environment is an open and timely question. This intervention will include two arms: the impact of the use of the mobile app for anxiety and for cancer related neuropathy.

ELIGIBILITY:
Inclusion Criteria

Anxiety Arm:

1. previous diagnosis of cancer, other than non-melanoma skin cancer
2. over 21 years of age
3. routine access to the Internet
4. comfortable reading and writing in English
5. have completed primary treatment for cancer
6. indicate the presence of cancer related anxiety as indicated by the PROMIS measure
7. not currently practicing meditation regularly (more than one hour per week), and
8. diagnosed with any stage of cancer
9. own a smartphone or tablet

Cancer Related Neuropathy Arm

1. diagnosis of cancer
2. use of a taxane or platinum agent
3. experiencing CIPN, per self-report
4. over 21 years of age
5. routine access to a smart device
6. comfortable reading and writing in English, and
7. not currently practicing meditation regularly (more than one hour per week).

Exclusion Criteria:

None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the impact of Mobile Mindful Meditation on anxiety as measured with the GAD-7 (Anxiety Arm) | 8 weeks
  Anxiety will be measured with the GAD-7, which entails respondents indicating how much in the past week they experienced anxiety. Participants are asked to provide their responses on a 5-point Likert type scale, with options ranging from "never" to "always."
Evaluate the impact of Mobile Mindful Meditation on pain as measured with the PEG-3 (Anxiety Arm) | 8 weeks
  Pain will be measured with the PEG-3, a three item measure assessing pain intensity, interference with general activity, and interference with enjoyment of life, with response options ranging from a 0-10 scale (0 being "no pain" or "does not interfere" and 10 being "pains as bad as you can imagine" or "completely interferes").
Evaluate the impact of Mobile Mindful Meditation on fatigue as measured with the Brief Fatigue Inventory (Anxiety Arm) | 8 weeks
  Fatigue will be measured with the Brief Fatigue Inventory, a 9-item measure where respondents are asked to rate their fatigue on an 11-point scale, with options on three items ranging from either "no fatigue" to "as bad as you can imagine" and options on the remaining items ranging from "does not interfere" to "completely interferes"
Evaluate the impact of Mobile Mindful Meditation on trauma as measured with the PCL-5 (Anxiety Arm) | 8 weeks
  Trauma Symptoms will be measured with the PCL-5. This 20-item measure assess for the 20 DSM-5 symptoms of PTSD, which fit into the larger categories of intrusive and avoidant symptoms.
Evaluate the impact of Mobile Mindful Meditation on sleep as measured by the PROMIS sleep scale (Anxiety Arm) | 8 weeks
  Sleep will be measured by the PROMIS sleep scale, an 8-item measure, with 5-point response choices.
Evaluate the impact of Mindfulness Coach on pain as measured with the McGill Pain Questionnaire (Neuropathy Arm) | 8 weeks
  This is a self-report questionnaire, consisting of 3 major classes of word descriptors--sensory, affective/emotional impact and cognitive evaluation of pain. The Short-form McGill Pain Questionnaire (SFMPQ) was developed to provide an instrument that could be completed in less time than the MPQ but would still reflect both the sensory and affective dimensions of pain and has been shown to have high correlations with the original McGill Pain Scale.
Evaluate the impact of Mindfulness Coach on anxiety as measured with the PROMIS anxiety (Neuropathy Arm) | Baseline, 8 weeks, 16 weeks
  This is a 22 item measure created for cancer survivors to measure both symptoms of anxiety and whether help was needed due to anxiety symptoms65. This is included at all time-points as an additional outcome measure.
Evaluate the impact of Mindfulness Coach on fatigue as measured with the BFI (Neuropathy Arm) | Baseline, 8 weeks, 16 weeks
  The Brief Fatigue Inventory (BFI) is a 15-item measure assessing both the severity of fatigue and the impact of fatigue on daily functioning64. This is included at all three time-points as an additional outcome measure.
Evaluate the impact of Mindfulness Coach on Quality of Life as measured with the FACT scale (Neuropathy Arm) | Baseline, 8 weeks, 16 weeks
  The FACT-GOC-Ntx scale includes 11 additional items (27 original items and 11 CIPN items) to measure the severity and impact of chemotherapy induced peripheral neuropathy. This data will serve as both a screening tool and baseline measure of CIPN.

SECONDARY OUTCOMES:
Evaluate the satisfaction with Mobile Mindfulness Meditation as measured by questionnaires on the Online Mindful Meditation platforms (Anxiety Arm) | Baseline, 16 weeks
  Patient self-reporting through the Mobile Mindful Meditation platform will measure satisfaction via the Five Facet Mindfulness Questionnaire. Successfully completing the 8-week program will also be an indirect measure of patient satisfaction.
Evaluate the satisfaction with Mindfulness Coach | Baseline, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erin O Bantum, PhD, Principal Investigator — University of Hawaii Cancer Research Center
Locations (2):
- United States (2):
  - Palo Alto VA Health Care System, Palo Alto, California
  - University of Hawaii Cancer Center, Honolulu, Hawaii

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orasud AS, Uchiyama M, Pagano I, Bantum E. Mobile Mindfulness Meditation for Cancer-Related Anxiety and Neuropathy: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 12;13:e47745. doi: 10.2196/47745. PMID 38345843